CLINICAL TRIAL: NCT01026506
Title: Pilot Study on the Effects of Oral Intervention With c9,t11-conjugated Linoleic Acid in Children and Adolescents With Allergic Asthma
Brief Title: c9,t11-CLA in Children and Adolescents With Allergic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: Cognis Deutschland GmbH & Co. KG (Industry)
Responsible Party: Prof. Dr. G. Jahreis, University of Jena, Dept. of Nutritional Physiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSEP H34-08
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Allergic Bronchial Asthma
Keywords: c9,t11-CLA; allergic bronchial asthma; children and adolescents
MeSH Terms: interventions — Linoleic Acids, Conjugated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: conjugated linoleic acid — 3 g/d of an esterified CLA preparation free of t10,c12-CLA (75% c9,t11-CLA, 87% purity) or placebo oil mixed in yoghurt for 12 weeks

SUMMARY:
The study was performed to investigate the effects of a dietary intervention with c9,t11-CLA on clinical and immunological parameters in children and adolescents with allergic bronchial asthma.

DETAILED DESCRIPTION:
In-vitro and animal studies strongly suggest that c9,t11-CLA reduces inflammatory processes in asthma-models. Aim of this study was to determine possible beneficial effects of orally administered c9,t11-CLA in children and adolescents with allergic bronchial asthma.

Thirty subjects (14 girls, 16 boys, age 6-18 years) were recruited from regular patients in the Clinic for Pediatric Allergology of the Friedrich Schiller University Jena. Informed consent was obtained from all participants/parents. 29 subjects completed the study.

The study was designed as a randomized and placebo-controlled study. After a 1-week run-in period to ascertain the current state of disease and categorization of allergic sensitization by RAST, the participants were randomized and evenly distributed to receive either 3 g/d of an esterified CLA preparation free of t10,c12-CLA (75% c9,t11-CLA, 87% purity) or 3 g/d of a placebo oil mixed in 100 g portions of milk fat-free yoghurt for 12 weeks. The yoghurt was freshly prepared and distributed in frequent intervals.

At the beginning and at the end of the study, lung function parameters were assessed by whole body plethysmography, and venous blood and 24h-urine samples were collected for further analyses. Throughout the entire study, the participants daily recorded their peak-flow data and kept protocol about their symptoms and drug usage.

ELIGIBILITY:
Inclusion Criteria:

* age 6-18 years
* doctor-diagnosed bronchial asthma
* allergic sensitization (house dust mite, grass pollen)
* willingness to use only the recommended drugs
* competence regarding the daily documentation of peak-flow data and symptoms

Exclusion Criteria:

* SIT within the last 2 years
* primary and secondary immune deficiency
* usage of systemic corticoids
* intolerance against milk protein
* alcohol and drug abuse

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
lung function parameters | 12 weeks

SECONDARY OUTCOMES:
symptom score, serum ECP, ex-vivo and in-vitro cytokine production of PBMC, urinary oxidation parameters, fatty acid distribution in erythrocytes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — University of Jena, Dept. of Nutritional Physiology
Locations (1):
- University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Jaudszus A, Mainz JG, Pittag S, Dornaus S, Dopfer C, Roth A, Jahreis G. Effects of a dietary intervention with conjugated linoleic acid on immunological and metabolic parameters in children and adolescents with allergic asthma--a placebo-controlled pilot trial. Lipids Health Dis. 2016 Feb 3;15:21. doi: 10.1186/s12944-016-0187-6. PMID 26843092